CLINICAL TRIAL: NCT00829296
Title: The Effects of Nebivolol on Aortic Impedance Parameters in Type 2 Diabetics
Brief Title: Safety Study to Lower the Risk of Heart Failure is Also Effective in Reducing Stiffness of the Arteries
Acronym: EFFORT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16310B (EFFORT trial); NCT01059916 (obsolete NCT alias)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension; Diabetes
Keywords: diabetes; hypertension; aortic impedance
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nebivolol (Experimental): Starting at dose of 5 mg daily titrated up to max of 40 mg until target BP of 130/80 is reached
  Interventions: Drug: nebivolol
- Metoprolol (Active Comparator): Starting at 50 mg daily dose is titrated to max 200 mg until target BP of 130/80 is reached
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: nebivolol — Starting at dose of 5 mg daily titrated up to max of 40 mg until target BP of 130/80 is reached
  Other Names: bystolic
  Arms: nebivolol
Drug: Metoprolol — Starting at 50 mg daily dose is titrated to max 200 mg until target BP of 130/80 is reached
  Other Names: lopressor
  Arms: Metoprolol

SUMMARY:
The study is being done to see if a drug shown to lower the risk of heart failure is also effective in reducing the stiffness of the arteries.

DETAILED DESCRIPTION:
To determine the effect of nebivolol versus metoprolol in Type 2 hypertensive diabetic patients on systolic blood pressure and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Established Type 2 diabetic not treated with insulin
* Stage 1 hypertensives blood pressure > 130/80 mmHg and < 160/100 mmHg
* BMI < 35
* Hemoglobin A1C < 8.5
* Must be postmenopausal or taking some form of birth control of surgically sterile

Exclusion Criteria:

* Acute myocardial infarction, unstable angina, stroke or TIA within the past year.
* Active angina in the last three months
* Diabetes requiring treatment with insulin
* Severe asthma
* Female who are pregnant, planning to be pregnant during the study period, lactating or women of childbearing potential who are not using a medically approved method of contraception
* Recent history of substance or alcohol abuse .
* Uncontrolled hypertension systolic blood pressure >160mmHg or diastolic blood pressure > 100 mmHg

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nebivolol: Starting at dose of 5 mg daily titrated up to max of 40 mg until target BP of 130/80 is reached
  nebivolol
- Metoprolol: Starting at 50 mg daily dose is titrated to max 200 mg until target BP of 130/80 is reached
  Metoprolol
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol
Started | 34 | 36
Completed | 29 | 32
Not Completed | 5 | 4
Not completed — Adverse Event | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (6.9) | 64.1 (6.1) | 64.5 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Systolic Blood Pressure (SBP)
Description: Changes in aortic impedance in patients on nebivolol vs. metoprolol succinate in Type 2 hypertensive diabetic patients as measured by the change from baseline in central systolic blood pressure.
Time Frame: Baseline and 26 Weeks
Population: Nine patients (4 in the Metoprolol and 5 in the Nebivolol group) discontinued the study medications early in the 26-week follow-up and did not undergo final assessment. Given that our interest was on efficacy, thus, results were reported only on those 61 patients (32 in the Metoprolol and 29 in the Nebivolol group) who completed the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 29 | 32
mmHg
  Aortic Systolic Blood Pressure at Baseline | 125.3 (8.0) | 127.8 (8.8)
  Aortic Systolic Blood Pressure at 26 Weeks | 121.6 (8.2) | 123.8 (11.1)

2. Secondary Outcome: Change in Pulse Wave Velocity (PWV)
Description: To examine the effect of nebivolol versus metoprolol succinate in Type 2 hypertensive diabetic patients on other measures of central conduit artery function such as pulse wave velocity.
Time Frame: Baseline and 26 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 29 | 32
m/s
  Pulse wave velocity at Baseline | 6.48 (0.8) | 6.52 (1.2)
  Pulse wave velocity at 26 Weeks | 6.3 (0.9) | 6.4 (1.3)

3. Secondary Outcome: Change in Augmentation Index
Description: Augmentation index is defined as the percentage of the central pulse pressure which is attributed to the reflected pulse wave and, therefore, reflects the degree to which central arterial pressure is augmented by wave reflection.
Time Frame: Baseline and 26 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 29 | 32
percent (%)
  Augmentation index at Baseline | 22.0 (7.1) | 26.2 (8.3)
  Augmentation index at 26 Weeks | 22.1 (7.4) | 24.6 (6.7)

4. Secondary Outcome: Change in Pulse Pressure Amplification
Description: To examine the effect of nebivolol versus metoprolol succinate in Type 2 hypertensive diabetic patients on other measures of central conduit artery function such as pulse pressure amplification (central pulse pressure /brachial pulse pressure).
Time Frame: Baseline and 26 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 29 | 32
ratio
  Pulse pressure amplification at Baseline | 0.77 (0.08) | 0.79 (0.09)
  Pulse pressure amplification at 26 Weeks | 0.83 (0.09) | 0.85 (0.12)

ADVERSE EVENTS:
Arm/Group | Nebivolol | Metoprolol
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 8/34 | 9/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=34) | Metoprolol (N=36)
Fatigue (General disorders) | 2 | 6
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dizziness (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No